CLINICAL TRIAL: NCT03389984
Title: Characterization of the Initial Psoriatic Skin Transcriptionnl Profile Associated to a Response to Adalimumab Therapy
Brief Title: Psoriatic Inflammation Markers Predictive of Response to Adalimumab
Acronym: IMPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMPRA
Record Dates: First submitted 2017-12-06; First posted 2018-01-04 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Diagnostic Test: cutaneous

INTERVENTIONS:
Diagnostic Test: cutaneous — SKIN BIOPSY

SUMMARY:
The objective is to compare the initial skin inflammatory transcriptomic profile of psoriatic patient responder to Adalimumab therapy (defined as the achievement of a Psoriasis Area and Severity Index 75 response at 16 weeks) with the transcriptomic profile of patient non-responder to Adalimumab therapy (defined as the non-achievement of a Psoriasis Area and Severity Index 50 response at 16 weeks) to identify differentially expressed genes in order to define predictive markers of response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque psoriasis involving at least 10% of body surface area, with a PASI score >10,
* Negative pregnancy test for women of childbearing potential, and use of an effective method of contraception,
* Pretreatment assessment to identify contraindications to anti-tumor necrosis factor-alpha therapy (chest x-ray and Intradermal reaction (detection of latent tuberculosis),
* Anti-tumor necrosis factor-alpha treatment with adalimumab has been prescribed

Exclusion Criteria:

* Classical exclusion criteria for adalimumab therapy (hypersensitivity to the product, severe heart failure, abscess, tuberculosis or other opportunistic infection),
* History of demyelinating disease, any unstable medical condition, patients with recurrent serious infections , history of cardiovascular or cerebrovascular disease , history of cancer
* Patients not having tuberculosis prophylaxis as per local guidelines for latent tuberculosis, or patients non-treated active tuberculosis
* Ongoing pregnancy or breastfeeding
* Absence of written consent,
* Prior treatment with one of the following anti-psoriatic treatments: biologics during the 3 months prior baseline visit, other systemic treatment during the 4 weeks prior baseline visit or topical therapy during the 2 weeks prior baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline messenger ribonucleic acid expression at 16 weeks of treatment | From baseline to 16 weeks treatment
  messenger ribonucleic acid expression assessed by quantitative reverse transcription-polymerase chain reaction

SECONDARY OUTCOMES:
Change from baseline drug and anti-drug concentrations at 16 weeks of treatment | From baseline to 16 weeks treatment
  assessed by enzyme-linked-immunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France